CLINICAL TRIAL: NCT03663829
Title: Impact of Anti-citrullinated Protein Antibody Status on Treatment Response and Treatment Persistence in Patients With Rheumatoid Arthritis Who Are Treated With Abatacept or Tumour Necrosis Factor Inhibitors. An Analysis From the Optimising Patient Outcome in Australian Rheumatology (OPAL) Registry.
Brief Title: Impact of Anti-citrullinated Protein Antibody Status on Treatment Response and Treatment Persistence in Participants With Rheumatoid Arthritis (RA) Who Are Treated With Abatacept or Tumor Necrosis Factor Inhibitors in Australia
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-728
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants RA who have received a TNFi
  Interventions: Other: Non-Interventional
- Participants with RA who have received abatacept
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional
  Groups: Participants RA who have received a TNFi
Other: Non-Interventional — Non-Interventional
  Groups: Participants with RA who have received abatacept

SUMMARY:
An observational study assessing the impact of anti-citrullinated antibody (ACPA) in rheumatoid arthritis (RA) participants who have received abatacept or tumour necrosis factor inhibitors (TNFi) from the Optimising Patient outcome in Australian rheumatoLogy (OPAL) registry

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis
* Have a baseline ACPA recorded
* Received either abatacept or a TNFi (adalimumab, certolizumab, etanercept or golimumab) during the sample selection window 1 August 2006 to 30 June 2017

Exclusion Criteria:

* Patients who have died
* Patients with concomitant inflammatory diseases (e.g. ankylosing spondylitis, psoriatic arthritis, Crohn's disease, ulcerative colitis)
* Patients who have no visit data recorded (even if medication data is available)

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of rheumatoid arthritis (RA) who have received a TNFi or abatacept and registered in the OPAL registry
Sampling Method: Probability Sample
Enrollment: 2052 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
ACPA (Anti-cyclic citrullinated peptide) status | Pre-Index
  ACPA-positive greater than or equal to 5 Ru/mL in Australia, greater than or equal to 20 Ru/mL in US

SECONDARY OUTCOMES:
Number of participants with positive ACPA | Index
  ACPA-positive greater than or equal to 5 Ru/mL in Australia, greater than or equal to 20 Ru/mL in US
Number of participants with negative ACPA | Index
  ACPA-negative less than or equal to 5 Ru/mL in Australia, less than or equal to 20 Ru/mL in US
CDAI (clinical disease activity index) score | Index plus or minus 1 month
  Remission CDAI <2.9 Low disease activity CDAI ≥ 2.9 but <10.0 Moderate disease activity CDAI ≥ 10.1 but <22.0 High disease activity CDAI ≥ 22.0
CDAI (clinical disease activity index) score | 12 months plus or minus 3 months
  Remission CDAI <2.9 Low disease activity CDAI ≥ 2.9 but <10.0 Moderate disease activity CDAI ≥ 10.1 but <22.0 High disease activity CDAI ≥ 22.0
DAS28 (disease activity score 28)-CRP-3 (C reactive protein) score | Index plus or minus 1 month
  The DAS-28 CRP-3 is a measure of disease activity in rheumatoid arthritis (RA) that assesses 28 joints in RA commonly affected. The DAS-28 CRP 3 takes into account tender and swollen joint counts and CRP level (measure of inflammation in the blood). The DAS-28 CRP 3 measure does not include patient global assessment of health.
DAS28 (disease activity score 28)-CRP-3 (C reactive protein) score | 12 months plus or minus 3 months
  The DAS-28 CRP-3 is a measure of disease activity in rheumatoid arthritis (RA) that assesses 28 joints in RA commonly affected. The DAS-28 CRP 3 takes into account tender and swollen joint counts and CRP level (measure of inflammation in the blood). The DAS-28 CRP 3 measure does not include patient global assessment of health.
Number of participants with treatment persistence | Approximately 11 years and 5 months
Number of participants with treatment discontinuation | Approximately 11 years and 5 months
Number of participants identified as taking abatacept | Index
Number of participants identified as taking TNFi (tumor necrosis factor inhibitor) | Index
Number of participants that achieved remission | 12 months plus or minus 3 months
  Remission CDAI <2.9 Low disease activity CDAI ≥ 2.9 but <10.0 Moderate disease activity CDAI ≥ 10.1 but <22.0 High disease activity CDAI ≥ 22.0

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Canberra City, Australia

REFERENCES:
- See also: BMS (Bristol-Myers Squibb) Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm